CLINICAL TRIAL: NCT03984630
Title: Feasibility of a Single Goal Intervention to Promote Appropriate Gestational Weight Gain
Brief Title: Pregnancy Intervention Revolving Around Goal-focused Education (GIRAFE)
Acronym: GIRAFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY0004032
Record Dates: First submitted 2019-06-10; First posted 2019-06-13 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Pregnancy
Keywords: Dietary Fiber; Gestational weight gain
MeSH Terms: conditions — Gestational Weight Gain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (No Intervention): Participants were informed to continue to receive usual care by their Obstetrician and were asked to send in body weights weekly.
- Intervention Arm (Experimental): Received snacks high in fiber, attended weekly phone calls, recorded daily food intake and reported weekly body weight for 12 weeks.
  Interventions: Behavioral: Dietary Fiber Intervention

INTERVENTIONS:
Behavioral: Dietary Fiber Intervention — Intervention included weekly group-based phone counseling with a Registered Dietitian (RD) to encourage consumption of a high fiber diet (≥30 g/day). All women reported their body weight weekly.
  Arms: Intervention Arm

SUMMARY:
The purpose of study is to learn if consuming ≥30 grams or more of fiber per day can help pregnant women gain an appropriate amount of weight during their pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Women between 9 to 15 weeks pregnant
* BMI between 22.0 - 40.0 kg/m2 and between the
* Ages of 18-45 years
* Able to be recruited from the University of Kansas Medical Center (KUMC).

Exclusion Criteria:

* No Internet access
* Consuming more than 20 grams per day of fiber
* And/or with the following medical conditions during pregnancy:
* Pre-gestational diabetes
* Diagnosed with diabetes
* Pre-eclampsia
* Hypertension
* Other metabolic abnormalities
* Asthma
* Heart disease
* Smoking
* Drug abuse
* Pregnancies of multiples

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2016-08-11 (Actual); Primary Completion 2017-02-09 (Actual); Study Completion 2017-04-20 (Actual)

PRIMARY OUTCOMES:
Proportion of excessive gestational weight gain based on weight gain guidelines. | 12-24 weeks gestation and during pregnancy

SECONDARY OUTCOMES:
Total gestational weight gain | 12-24 weeks gestation and during pregnancy
  Measure gestational weight gain (kg) for those women in the intervention arm and control arm.
Total dietary fiber intake | 12-24 weeks gestation and during pregnancy
  ≥30 g/day

CONTACTS AND LOCATIONS:
Overall Officials: Holly Hull, PhD, Principal Investigator — University of Kansas Medical Center

REFERENCES:
- [Derived] Hull HR, Herman A, Gibbs H, Gajewski B, Krase K, Carlson SE, Sullivan DK, Goetz J. The effect of high dietary fiber intake on gestational weight gain, fat accrual, and postpartum weight retention: a randomized clinical trial. BMC Pregnancy Childbirth. 2020 May 24;20(1):319. doi: 10.1186/s12884-020-03016-5. PMID 32448177